CLINICAL TRIAL: NCT02383576
Title: Retrospective Data Collection: Post Study Treatment Anticancer Therapy From All Randomized Patients Involved in IMELDA MO22223
Brief Title: Retrospective Data Collection: Post Study Treatment Anticancer Therapy From IMELDA MO22223
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: MO29587
Record Dates: First submitted 2015-03-04; First posted 2015-03-09 (Estimated); Results first posted 2018-04-13 (Actual); Last update posted 2018-04-13 (Actual); Status verified 2017-09

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Bevacizumab: Participants who received bevacizumab in IMELDA (MO22223) P-trial and were in maintenance phase were observed.
  Interventions: Other: No Intervention
- Bevacizumab and Capecitabine: Participants who received bevacizumab and capecitabine in IMELDA (MO22223) P-trial and were in maintenance phase were observed.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — No intervention administered in this study.

SUMMARY:
This study aims to understand better the effective results from the IMELDA MO22223 P-trial (NCT00929240) and see if the anti-cancer therapies given during its follow-up time after study treatments were terminated possibly had an effect on efficacy results.

ELIGIBILITY:
Inclusion Criteria:

Having been randomized in the IMELDA MO22223 P-trial

Exclusion Criteria:

Not having been randomized in the IMELDA MO22223 P-trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All participants randomized in IMELDA (MO22223)
Sampling Method: Probability Sample
Enrollment: 185 (Actual)
Dates: Start 2015-04-30 (Actual); Primary Completion 2016-01-22 (Actual); Study Completion 2016-01-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Reference Study ID Number: MO29587 www.roche.com/about_rouche/roche_worldwide.htm, Study Director — Hoffmann-La Roche
Locations (32):
- Brazil (8):
  - Crio - Centro Regional Integrado de Oncologia, Fortaleza, Ceará
  - Instituto Nacional de Cancer - INCa; Oncologia, Rio de Janeiro, Rio de Janeiro
  - Hospital de Caridade de Ijui; Oncologia, Ijuí, Rio Grande do Sul
  - Hospital das Clinicas - UFRGS, Porto Alegre, Rio Grande do Sul
  - Hospital Amaral Carvalho, Jaú, São Paulo
  - Faculdade de Medicina do ABC - FMABC; Oncologia e Hematologia, Santo André, São Paulo
  - Instituto do Cancer do Estado de Sao Paulo - ICESP, São Paulo, São Paulo
  - Hospital Santa Marcelina;Oncologia, São Paulo, São Paulo
- France (8):
  - HOPITAL JEAN MINJOZ; Oncologie, Besançon
  - Chg de Chartres Hopital Louis Pasteur; Pneumologie, Chartres
  - Clinique Sainte Marguerite; Oncologie Medicale, Hyères
  - Centre Bourgogne, Service de Radiotherapie, Lille
  - Institut Curie; Oncologie Medicale, Paris
  - HOPITAL TENON; Cancerologie Medicale, Paris
  - Clinique Francheville; Radiotherapie, Périgueux
  - Institut D Oncologie Medical, Strasbourg
- India (2):
  - Tata Memorial Hospital; Dept of Medical Oncology, Mumbai, Maharashtra
  - Rajiv Gandhi Cancer Inst.&Research Center; Medical Oncology, New Delhi, National Capital Territory of Delhi
- Italy (3):
  - Ospedale Antonio Perrino; Oncologia Medica, Brindisi, Apulia
  - Università Federico II; Dip. Di Endocrinologia ed Oncologia Molecolare e Clinica, Napoli, Campania
  - Uni Degli Studi Di Genova ; Clinica Di Medicina Interna Ad Indirizzo Oncologico, Genoa, Liguria
- Spain (8):
  - Hospital Virgen de los Lirios; Servicio de Oncologia, Alcoy, Alicante
  - Corporacio Sanitaria Parc Tauli; Servicio de Oncologia, Sabadell, Barcelona
  - Complejo Hospitalario la Mancha Centro;Servicio Oncologia, Alcazar de S. Juan, Ciudad Real
  - Hospital de Cruces; Servicio de Oncologia, Barakaldo, Vizcaya
  - Complejo Hospitalario de Jaen-Hospital Universitario Medico Quirurgico; Servicio de Oncologia, Jaén
  - Hospital Clinico Universitario Virgen de la Victoria; Servicio de Oncologia, Málaga
  - Complejo Hospitalario de Toledo- H. Virgen de la Salud; Servicio de Oncologia, Toledo
  - Hospital Universitario la Fe; Servicio de Oncologia, Valencia
- Turkey (Türkiye) (3):
  - Gazi Uni Medical Faculty Hospital; Oncology Dept, Ankara
  - Akdeniz University Medical Faculty; Medical Oncology Department, Antalya
  - Hacettepe Uni Medical Faculty Hospital; Oncology Dept, Sıhhiye, Ankara

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bevacizumab | Bevacizumab and Capecitabine
Started | 94 | 91
Completed | 31 | 46
Not Completed | 63 | 45
Not completed — Death | 53 | 33
Not completed — Lost to Follow-up | 7 | 1
Not completed — Withdrew Consent | 1 | 6
Not completed — Investigator's Decision | 0 | 1
Not completed — Administrative/Other | 2 | 4

BASELINE CHARACTERISTICS:
Population: It is a retrospective collection of additional anti-cancer medications that participants might have taken after a progression free survival (PFS) event in the main Imelda study. Demographic data was not collected.
Groups:
- Total: Total of all reporting groups
Arm/Group | Bevacizumab | Bevacizumab and Capecitabine | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Continuous [unit: years]
Sex: Female, Male

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Prematurely Withdrawn From Maintenance Therapy
Description: Participants who had prematurely withdrawn from maintenance study treatment were reported. The retrospectively collected data was pooled with the data collected within the IMELDA (MO22223) P-trial to allow a statistically meaningful analysis.
Time Frame: Up to 78 months
Population: The main analysis population was based on those participants of the maintenance phase Intent-to-Treat population (ITT) population (all randomized participants) of the IMELDA (MO22223) P-trial, who had consented to participate in this follow-up study.
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab | Bevacizumab and Capecitabine
Number analyzed (Participants) | 59 | 59
percentage of participants | 93.2 | 84.7

2. Primary Outcome: Percentage of Participants Who Received Further Anti-Cancer Therapies After Discontinuation of Study Treatment
Description: Participants who received further anti-cancer therapies after discontinuation of study treatment were reported. The retrospectively collected data was pooled with the data collected within the IMELDA (MO22223) P-trial to allow a statistically meaningful analysis.
Time Frame: Up to 78 months
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab | Bevacizumab and Capecitabine
Number analyzed (Participants) | 59 | 59
percentage of participants | 94.9 | 91.5

3. Primary Outcome: Time From Last Maintenance Study Medication Start to Start of Further Anti-Cancer Therapy
Description: Time from last maintenance study medication to the start of any further anti-cancer therapy was reported. The retrospectively collected data was pooled with the data collected within the IMELDA (MO22223) P-trial to allow a statistically meaningful analysis.
Time Frame: Up to 78 months
Population: as for outcome 1
Measure: Median (Full Range); unit: days
Arm/Group | Bevacizumab | Bevacizumab and Capecitabine
Number analyzed (Participants) | 59 | 59
days | 22.5 [0 to 70] | 23.5 [0 to 630]

4. Primary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as the time from start of the study to the first documented occurrence of disease progression. The retrospectively collected data was pooled with the data collected within the IMELDA (MO22223) P-trial to allow a statistically meaningful analysis.
Time Frame: Up to 78 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab | Bevacizumab and Capecitabine
Number analyzed (Participants) | 59 | 59
months | 4.3 [2.7 to 6.8] | 12.2 [7.6 to 15.4]

5. Primary Outcome: Overall Survival
Description: Overall survival was defined as the interval between start of the study and the date of death from any cause. The retrospectively collected data was pooled with the data collected within the IMELDA (MO22223) P-trial to allow a statistically meaningful analysis.
Time Frame: Up to 78 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab | Bevacizumab and Capecitabine
Number analyzed (Participants) | 59 | 59
months | 22.3 [12.1 to 29.8] | 36.5 [27.6 to NA] — Upper limit of 95% CI was not reached.

ADVERSE EVENTS:
Description: This study only collected retrospective data on anti-cancer therapies taken by patients after the end of the IMELDA (MO22223) P-trial and no adverse event data was collected in this study.
Arm/Group | Bevacizumab | Bevacizumab and Capecitabine
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.